CLINICAL TRIAL: NCT00816790
Title: A Comparison of Standard Vs Renal Dosing of Piperacillin/Tazobactam in Acute Renal Failure and Septic Shock
Brief Title: Standard Vs Adjusted Dosing of Piperacillin/Tazobactam in Acute Renal Failure and Septic Shock
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped because of study personel movement to another institution.
Sponsor: Fraser Health (Other)
Responsible Party: Principal Investigator, Sean Keenan, Intensivist, Fraser Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FHREB 2008-085
Record Dates: First submitted 2008-12-31; First posted 2009-01-05 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Septic Shock; Acute Renal Failure
Keywords: Septic shock; Acute Renal Failure; Antimicrobial; Drug Dosing; Feasibility Study
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury | interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Adjusted (Active Comparator): This arm will receive their broad spectrum antibiotic as an adjusted dose based on their renal function as measured when sepsis is diagnosed and antimicrobials are initiated
  Interventions: Drug: Piperacillin/Tazobactam
- Unadjusted Dose (Experimental): This arm will receive their broad spectrum antibiotic as an unadjusted dose regardless of their renal function
  Interventions: Drug: Piperacillin/Tazobactam

INTERVENTIONS:
Drug: Piperacillin/Tazobactam — eGFR 20-40 mls/min: Piperacillin/Tazobactam 3.375g IV q6h x 24 hours eGFR < 20 mls/min: Piperacillin/Tazobactam 2.25g IV q6h x 24 hours
  Other Names: Tazocin
  Arms: Dose Adjusted
Drug: Piperacillin/Tazobactam — Piperacillin/Tazobactam 4.5g IV q 6h x 24 hours
  Other Names: Tazocin
  Arms: Unadjusted Dose

SUMMARY:
The objective of this study is to determine the feasibility of conducting a large scale randomized controlled trial comparing standard and renally adjusted dosage of antibiotics in the septic shock patients with acute renal dysfunction. We will use Piperacillin as the prototype antibiotic in our study.

DETAILED DESCRIPTION:
Septic shock is a significant cause of morbidity and mortality. Early Goal Directed therapy, fluid resuscitation, use of vasopressors and/or inotropes, and appropriate empiric antibiotic administration remain the cornerstone of therapy in the treatment of septic shock. Despite aggressive interventions, the death rate from septic shock in North America remains as high as 50 percent.

Septic shock is defined as severe sepsis with hypotension not reversed by adequate fluid resuscitation. This state of distributive shock often results in hypo-perfusion of all major organ systems, including the kidneys, and is a common cause of multi-organ failure. Acute renal failure in the setting of septic shock often leads clinicians to adjust dosing of empiric antibiotics according to the apparent renal function. Renally adjusted antibiotic dosing in septic shock may be insufficient for several reasons. First, renal failure secondary to hypoperfusion often reverses following fluid resuscitation and vasopressor use, leading to subsequent under dosing. Second, a hypoperfusion state theoretically results in a reduction in the amount of antibiotic delivered to the site of infection. Lastly, for drugs with large volumes of distribution or prolonged half lives, large initial doses are required to quickly to achieve therapeutic concentrations.

To date, no studies have attempted to answer this important question by comparing standard doses to renally adjusted doses of empiric antibiotics in patients with both septic shock and renal dysfunction during the initial resuscitative period. Currently there is no uniform practice among clinicians with respect to antibiotic dosing, which reflects the paucity of evidence in this area. Some clinicians currently use full dosing of antibiotics in the setting of septic shock with acute renal failure while others adjust the dose based on renal function. Well designed, prospective, randomized controlled trials are urgently needed to clarify the role of antibiotic adjustment during the resuscitative period of septic shock.

The objective of this study is to determine the feasibility of conducting a large scale randomized controlled trial comparing standard and renally adjusted dosage of antibiotics in the septic shock patients with acute renal dysfunction. We will use Tazocin as the prototype antibiotic in our study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with septic shock according to the Surviving Sepsis Campaign
* Age > 19
* Most recent eGFR<40 mls/min

Exclusion Criteria:

* Pregnant
* Known chronic renal failure patients who are dialysis dependant
* Administration of systemic antibiotics > 1 dose
* Not expected to survive 28 days due to an underlying medical illness
* Allergy to Piperacillin/Tazobactam or any components of formulation within

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To determine rate of patient accrual (ability to identify and enrol patients in a timely fashion) and protocol adherence for this pilot randomized controlled trial. | 4 months

SECONDARY OUTCOMES:
ICU and hospital mortality. ICU and hospital length of stay. Duration of mechanical ventilation. | 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Sean Keenan, MD, Principal Investigator — Fraser Health Authority; Matthew Wiens, BSc PharmD, Study Director — Fraser Health Authority; Vincent Mabasa, BSc PharmD, Study Director — Fraser Health Authority; Sanjiv Kangura, BSc, Study Director — Fraser Health Authority
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada